CLINICAL TRIAL: NCT02189109
Title: A Phase 1b Dose-finding, Pharmacokinetic and Pharmacodynamic Study of NVX-108 Combined With Radiation and Temozolomide in Patients With Newly-diagnosed Glioblastoma Multiforme
Brief Title: The Effects of NVX-108 as a Radiation Sensitizer in Glioblastoma
Acronym: GBM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NuvOx LLC (Industry)
Collaborators: The Alfred (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVX108-GBM1B
Record Dates: First submitted 2014-05-19; First posted 2014-07-14 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Glioblastoma Multiforme
Keywords: glioblastoma; multiforme; radiation; radiation therapy
MeSH Terms: conditions — Glioblastoma | interventions — perfluoropentane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation (Experimental): NVX-108 (DDFP liquid emulsion) i.v. in conjunction with Radiation Treatment and Temozolimide. 0.05-0.35cc/kg.
  Interventions: Drug: NVX-108

INTERVENTIONS:
Drug: NVX-108 — 0.2% emulsion administered i.v.
  Other Names: Dodecafluoropentane

SUMMARY:
This clinical trial is testing the safety, tolerability and effectiveness of NVX-108 administered via intravenous infusion in combination with standard radiation and chemotherapy.

NVX-108 is being developed to increase the amount of oxygen delivered to tumors which is hoped to increase the effectiveness of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed newly-diagnosed glioblastoma multiforme.
2. No prior treatment for glioblastoma apart from surgical resection.
3. No prior treatment for glioblastoma apart from surgical resection.
4. Planned for 60 Gray of focal radiation administered in 30 fractions, concurrently with temozolomide chemotherapy.
5. Manageable risks associated with potential radiation necrosis in the radiation field, based on size of the field and proximity to eloquent brain regions (as assessed by the investigator).
6. Aged 18-70 years.
7. ECOG performance status 0-2.
8. Life expectancy of at least 3 months.
9. If receiving glucocorticoid therapy, the dose must be stable over at least 7 days prior to study enrollment.
10. Archived tumor tissue available for central review.
11. Able to undergo gadolinium-enhanced MRI (Gd-MRI) scans.
12. Baseline MRI performed within 14 days before starting study treatment, while on a stable glucocorticoid dose for at least 5 days before and during the imaging study.
13. Adequate hematologic, renal and hepatic function, as defined by:

    Absolute neutrophil count (ANC) ≥ 1.5 109/L Platelet count ≥ 100 109/L Hemoglobin ≥ 90 g/L International normalized ratio (INR) and activated partial thromboplastin time (APTT) < 1.5 upper limit of normal (ULN) Plasma creatinine< 1.5 ULN Total bilirubin within normal limits (< 2.5 ULN if Gilbert's syndrome) AST and ALT < 2.5 ULN
14. Patients who are women of childbearing potential or men (unless vasectomised) must agree to use a highly-effective method of birth control, such as hormonal contraceptive implants, combined oral contraceptives, an intrauterine device, a double-barrier method (eg. condom with a diaphragm) or abstinence, from study entry until 4 months after completing study therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
15. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Presence of leptomeningeal disease or multifocal glioblastoma that cannot be encompassed within a feasible and safe radiation field.
2. Intracranial bleeding, except for stable grade 1 hemorrhage.
3. Has not recovered from the adverse effects of surgical resection or biopsy, except for neurological deficits.
4. Patients who have received any other investigational agent within 4 weeks before enrollment.
5. Stroke or transient ischemic attack within 6 months before enrollment.
6. Myocardial infarction within 6 months before enrollment, unstable angina, New York Heart Association class II or greater congestive heart failure, or uncontrolled hypertension (systolic BP > 160 mmHg and/or diastolic BP > 100 mmHg).
7. Congenital long QT syndrome.
8. Clinically-significant chronic obstructive pulmonary disease or asthma.
9. Active major infection requiring treatment.
10. A history of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer or other solid tumors curatively treated with no evidence of disease for ≥ 2 years.
11. Known infection with human immunodeficiency virus or hepatitis B or C virus.
12. Current anticoagulant or antiplatelet therapy, except for prophylactic doses of low molecular weight heparins or low-dose aspirin.
13. History of allergic reactions attributed to compounds of similar chemical composition to NVX-108.
14. Women who are pregnant or breast feeding.
15. Inability to comply with study procedures.
16. History or evidence of any other clinically-significant condition that, in the opinion of the investigator, would pose a risk to subject safety or interfere with study procedures, evaluation or completion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-05; Primary Completion 2017-08-31 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of NVX-108 in Combination with Radiation and Temozolomide Defined by no Drug related Adverse Events (AE) in No More than 1 Patient per Treatment Group | 6 months
  Adverse Events are considered to be neurological and hemodynamic

SECONDARY OUTCOMES:
Progression Free Survival at 6 months | 6 months

OTHER OUTCOMES:
Tumor Reduction Based on Gd-MRI | 4 months
  First determination will be measured at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MBBSPhDFRACP, Principal Investigator — Nucleus Network
Locations (4):
- Australia (4):
  - St. Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Flinders Medical Centre, Adelaide, South Australia
  - Nucleus Network, Melbourne, Victoria
  - Epworth Center, Melbourne, Victoria

REFERENCES:
- [Derived] Lickliter JD, Ruben J, Kichenadasse G, Jennens R, Gzell C, Mason RP, Zhou H, Becker J, Unger E, Stea B. Dodecafluoropentane Emulsion as a Radiosensitizer in Glioblastoma Multiforme. Cancer Res Commun. 2023 Aug 21;3(8):1607-1614. doi: 10.1158/2767-9764.CRC-22-0433. eCollection 2023 Aug. PMID 37609003